CLINICAL TRIAL: NCT00426868
Title: A Randomized Clinical Trial of adiPose-deRived stEm & Regenerative Cells In the Treatment of Patients With Non revaScularizable ischEmic Myocardium - The PRECISE Trial
Brief Title: A Randomized Clinical Trial of Adipose-derived Stem Cells in Treatment of Non Revascularizable Ischemic Myocardium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRECISE-01
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Heart Disease; Coronary Arteriosclerosis; Cardiovascular Disease; Coronary Disease; Coronary Artery Disease
Keywords: ADRC; Stem Cells; chronic ischemia; heart disease; coronary artery disease; inducible reversible ischemia
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Direct injection of ADRCs into the Left Ventricle
- Placebo (Placebo Comparator)
  Interventions: Other: Direct injection of placebo into the Left Ventricle

INTERVENTIONS:
Other: Direct injection of ADRCs into the Left Ventricle — Dose escalation
  Arms: Treatment
Other: Direct injection of placebo into the Left Ventricle
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish safety and feasibility of utilizing Adipose Derived Stem & Regenerative Cells (ADRCs) in patients who have areas of myocardium that are not revascularizable and have demonstrated reversible ischemia.

DETAILED DESCRIPTION:
Subjects who have coronary artery disease that cannot be revascularized and demonstrate reversible ischemia in the area supplied by the non-revascularizable vessel(s) will be evaluated for eligibility in this study. Eligible subjects will undergo standard pre-operative testing after admission to the hospital, and then will undergo liposuction under anesthesia, after which ADRCs will be isolated from the lipoaspirate. According to randomization subjects will receive either ADRCs or placebo.

The outcomes of this trial will be based on assessment of primary and secondary endpoints at 6 months post index procedure. Long Term Follow-up will be conducted at 12, 18, 24 and 36 months after the procedure.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide written informed consent
* Males or females 20 to 75 years of age, inclusive
* Coronary artery disease not amenable to any type of revascularization procedure (percutaneous or surgical) in the target area
* Hemodynamic stability
* Ability to undergo liposuction
* Ability to walk on a treadmill
* Negative urine pregnancy test (females only).

Key Exclusion Criteria:

* Unstable angina
* Serum creatinine >2.5 mg/dL
* Planned or scheduled staged treatment of CAD or other interventional or surgical procedures
* Cardiogenic shock
* History of resuscitated sudden cardiac death; or symptomatic or sustained ventricular fibrillation or ventricular tachycardia.
* Vascular anatomy that precludes cardiac catheterization
* Peripheral artery disease that precludes insertion of an 8 Fr sheath
* Severe valvular disease
* Pregnant or nursing females
* Known and relevant allergies or sensitivities
* Life expectancy <1 year
* Participation in any other clinical research study that has not reached its primary endpoint or otherwise would interfere with the subject's participation in this study
* Any concurrent disease or condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety - Determined by Major Adverse Cardiac and Cerebral Events (MACCE) | Up to 36 months

SECONDARY OUTCOMES:
Feasibility - Assessment of cardiac function using a variety of functional and imaging studies including MRI, SPECT and Echocardiography | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Milstein, MD, Study Director — Cytori Therapeutics, Inc; Francisco J Fernández-Avilés, MD, PhD, FACC, FESC, Principal Investigator — Hospital G.U. Gregorio Marañón; Emerson C Perin, MD, PhD, Principal Investigator — Texas Heart Institute
Locations (4):
- Rigshospitalet University Hospital, Copenhagen, Denmark
- Netherlands (2):
  - Erasmus University Medical Centrum, Thorax Center, Rotterdam
  - University of Utrecht Medical Center, Utrecht
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Perin EC, Sanz-Ruiz R, Sanchez PL, Lasso J, Perez-Cano R, Alonso-Farto JC, Perez-David E, Fernandez-Santos ME, Serruys PW, Duckers HJ, Kastrup J, Chamuleau S, Zheng Y, Silva GV, Willerson JT, Fernandez-Aviles F. Adipose-derived regenerative cells in patients with ischemic cardiomyopathy: The PRECISE Trial. Am Heart J. 2014 Jul;168(1):88-95.e2. doi: 10.1016/j.ahj.2014.03.022. Epub 2014 Apr 5. PMID 24952864